CLINICAL TRIAL: NCT02519595
Title: Optimal Dosing of Ketamine for Procedural Sedation and Analgesia in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Nirupama Kannikeswaran, Associate Professor of Pediatrics and Emergency Medicine, Children's Hospital of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1-2013-88
Record Dates: First submitted 2015-08-05; First posted 2015-08-11 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Moderate, Deep Sedation
Keywords: Procedural sedation; ketamine; children
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ketamine IV 1 mg/kg (Experimental): Intervention: A blinded dose of 1mg/kg IV ketamine is administered to patients
  Interventions: Drug: Ketamine IV 1mg/kg
- Ketamine IV 1.5 mg/kg (Experimental): Intervention: A blinded dose of 1.5mg/kg IV ketamine is administered to patients
  Interventions: Drug: Ketamine IV 1.5mg/kg
- Ketamine IV 2 mg/kg (Experimental): Intervention: A blinded dose of 2 mg/kg IV ketamine is administered to patients
  Interventions: Drug: Ketamine IV 2mg/kg

INTERVENTIONS:
Drug: Ketamine IV 1mg/kg — Intervention: Ketamine IV 1mg/kg
  Arms: ketamine IV 1 mg/kg
Drug: Ketamine IV 1.5mg/kg — Intervention: Ketamine IV 1.5 mg/kg
  Arms: Ketamine IV 1.5 mg/kg
Drug: Ketamine IV 2mg/kg — Intervention: Ketamine IV 2 mg/kg
  Arms: Ketamine IV 2 mg/kg

SUMMARY:
There is a wide variation of published IV ketamine dosing regimens used for procedural sedation in children in the Emergency Department (ED). The purpose of the study was to compare the efficacy, duration of sedation and adverse events between the three commonly administered doses of IV ketamine (1 mg/kg, 1.5 mg/kg and 2 mg/kg) using the traditional administration method of 30-60 second infusion for ED sedation in children.

DETAILED DESCRIPTION:
This was a prospective, double-blind, randomized controlled trial of children aged 3 to 18 years who received IV ketamine for procedural sedation and analgesia (PSA) for orthopedic procedures, incision and drainage (I & D) of skin abscess and laceration repair in an inner city, tertiary care pediatric ED. Random sequence allocation was performed using a computer-generated, random number table by the study research pharmacist. The study participants were grouped according to their age as follows (1) 3-6 years (2) 7-12 years (3) 13-18 years. Children from each age group were assigned in equal numbers to all three ketamine dosing (1 mg/kg, 1.5 mg/kg and 2 mg/kg) groups using random permuted blocks stratified by the pharmacist. All ED staff including the physician and the nurse in charge of sedation, the study research assistant, the parents/guardians and the study subjects were blinded to the randomization and the group assignments. The dosage and administration of additional doses of ketamine were left to the discretion of the ED physician in charge of the sedation. The research team did not participate in the clinical care including sedation of the patient. Children were monitored per ED policy for the entire duration of sedation. Three 1 ml blood samples for the ketamine assay was collected from the existing intravenous access at three time intervals: 3-5 minutes after ketamine administration, at midpoint during the procedure and prior to discharge of the patient from the ED. In the event a second dose of ketamine was administered, a 4th 1 ml sample was collected 3-5 minutes after the 2nd dose in children weighing >20 kilograms. Patient demographics, procedure type, NPO status , ASA classification, pain medication administered prior to sedation (timing, dosage and type), number and total doses of ketamine administered after the initial study dose, sedation efficacy and duration, length of procedure, adverse events related to sedation, interventions performed to address the adverse events and patient disposition were collected. The study research assistant also performed a follow up phone call to the parents/caregivers of the children 48 hours after ED discharge to collect information on adverse events that happened at home . A total of 3 attempts were made to contact the parent/caregiver after which the participant was considered as lost to followup.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 -18 years of age
* Belonging to American Society of Anesthesiologists (ASA) classification 1 or 2
* Receiving IV ketamine for procedural sedation for orthopedic procedures,
* Incision and Drainage of skin abscess and laceration repair

Exclusion Criteria:

* Contraindications to use of Ketamine
* Parents or legal guardian not available or declined to provide informed consent
* Child declined to provide assent,
* Patients that received intramuscular ketamine,
* Patient that received benzodiazepines in addition to ketamine
* Children weighing >100 kilogram
* Children with developmental disabilities.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at a level 1 trauma Pediatric Emergency Department from July 1st 2010 to August 31st 2012. We enrolled a convenience sample of eligible patients. Study participants were identified using the electronic medical tracking board which lists the presenting complaint and after need for IV ketamine sedation was established with physician.
Pre-assignment Details: 11 consented patients were excluded as sedation and procedure was performed in the operating room rather than in the Emergency Department
Period: Overall Study
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Started | 58 | 57 | 56
Completed | 50 | 35 | 40
Not Completed | 8 | 22 | 16
Not completed — Protocol Violation | 8 | 22 | 16

BASELINE CHARACTERISTICS:
Population: Children aged3-18 years who received procedural sedation and analgesia in the Emergency Department
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg | Total
Number analyzed (Participants) | 50 | 35 | 40 | 125
Age, Customized [Number; unit: participants]
  3-6 years | 22 | 18 | 16 | 56
  7-12 years | 22 | 13 | 18 | 53
  13-18 years | 6 | 4 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 13 | 54
  Male | 27 | 17 | 27 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 6 | 14
  Not Hispanic or Latino | 39 | 31 | 32 | 102
  Unknown or Not Reported | 4 | 3 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 27 | 18 | 66
  White | 16 | 5 | 11 | 32
  More than one race | 4 | 0 | 1 | 5
  Unknown or Not Reported | 6 | 3 | 9 | 18
AMerican Society of Anesthesiologists (ASA) Category [Number; unit: participants] — The purpose of the ASA is to evaluate the degree of a patient's "sickness" or "physical state" before selecting the sedative or before performing the procedure. There are 6 categories
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  6. A declared brain-dead person whose organs are being removed for donor purposes.
  participants
    ASA Class 1, A normal healthy patient | 50 | 32 | 37 | 119
    ASA class 2, Mild systemic disease | 0 | 2 | 3 | 5
    ASA class 3, Severe systemic disease | 0 | 1 | 0 | 1
Procedure Type [Number; unit: participants]
  Fracture/Dislocation Reduction | 33 | 21 | 35 | 89
  Incision and Drainage | 12 | 11 | 2 | 25
  Laceration Repair | 5 | 3 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Sedation Efficacy
Description: Measure sedation depth using Ramsay Sedation Scale. Varies from 1-6 with 1: anxious, agitated, restless 2: Cooperative, oriented, tranquil 3: responsive to commands 4: Brisk response to light glabellar tap or auditory stimulus 5: Sluggish response to light glabellar tap or loud auditory stimulus 6 being no response to light glabellar tap or loud auditory stimulus. Higher the score, greater is the depth of sedation. Use of ketamine usually provides a depth of sedation of 5 or 6.
Time Frame: Participants will be assessed after study drug adminsitration and the maximum depth of sedation achieved recorded. Approximately 2 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 50 | 35 | 40
units on a scale | 5.5 [4 to 6] | 6 [4 to 6] | 6 [5 to 6]
Statistical Analysis 1: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Test type: Superiority or Other; p = 0.2, Kruskal-Wallis

2. Primary Outcome: Pain
Description: Measure pain using self reported Wong Baker faces pain rating scale prior to sedation, during sedation and prior to discharge.The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst". The patient must choose the face that best describes how they are feeling. The score has values of 0(no hurt), 2(hurts little bit), 4(hurts little more), 6(hurts even more), 8(hurts whole lot),10 (hurts worst). The patient chooses one number that describes the pain best (eg. Either a 2 or 4).
Time Frame: Patients will be assessed during the procedure after administration of sedation medicaiton. Approximately 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 50 | 35 | 40
units on a scale | 0 [0 to 4] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Test type: Superiority or Other; p = 0.09, Kruskal-Wallis

3. Secondary Outcome: Sedation Duration
Description: Length of sedation was defined as the time duration from the administration of study medication until ready for discharge using standardized discharge criteria (Aldrete scoring >9) followed at our institution.
Time Frame: Patients will be assessed during the length of time from administration of sedation medication until ready for discharge, Approximately 3 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 50 | 35 | 40
Minutes | 23 [19 to 38] | 24.5 [17.5 to 34.5] | 23 [19 to 29]
Statistical Analysis 1: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Test type: Superiority or Other; p = 0.2, Kruskal-Wallis

4. Secondary Outcome: Additional Dose
Description: Number of participants to whom additional doses of ketamine administered apart from the study dose
Time Frame: Patients will be assessed during procedure . Approximately 1 hours
Measure: Number; unit: participants
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 50 | 35 | 40
participants | 8 | 1 | 2

5. Secondary Outcome: Adverse Events
Description: Adverse events secondary to sedation experienced by the patient and interventions performed to overcome them
Time Frame: Patients will be assessed after administration of medication until discharge and will have a follow up phone call 48 hours after discharge for 3 attempts. 5 days.,
Measure: Number; unit: participants
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 50 | 35 | 40
participants
  Adverse events in ED | 5 | 5 | 4
  Post discharge Emesis | 4 | 4 | 6
Statistical Analysis 1: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Adverse events in ED; Test type: Superiority or Other; p = 0.8, Chi-squared
Statistical Analysis 2: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Post discharge Emesis; Test type: Superiority or Other; p = 0.5, Chi-squared

6. Secondary Outcome: Sedation Satisfaction
Description: Consultants will be asked to rate their level of satisfaction with sedation on a Likert Scale of 1-3
Time Frame: At the end of the procedure. Approximately 1 hour
Population: consultant satisfaction missing in 6 participants
Measure: Number; unit: participants
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Number analyzed (Participants) | 49 | 34 | 36
participants
  Not satisfied | 10 | 2 | 1
  Satisfied | 12 | 3 | 6
  Very Satisfied | 27 | 29 | 29
Statistical Analysis 1: Comparison: Ketamine IV 1 mg/kg vs Ketamine IV 1.5 mg/kg vs Ketamine IV 2 mg/kg; Test type: Superiority or Other; p = 0.011, Chi-squared

ADVERSE EVENTS:
Arm/Group | Ketamine IV 1 mg/kg | Ketamine IV 1.5 mg/kg | Ketamine IV 2 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/35 | 0/40
Other Adverse Events (participants affected / at risk) | 5/50 | 5/35 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine IV 1 mg/kg (N=50) | Ketamine IV 1.5 mg/kg (N=35) | Ketamine IV 2 mg/kg (N=40)
Oxygen Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) — Pulse oximetry <90% in room air
Emesis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) — Vomiting during/post sedation
Unpleasant Recovery Reaction (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) — agitation, hallucinations
Others (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Rash

LIMITATIONS AND CAVEATS:
Convenience sample of patients enrolled. One fourth of patients did not receive the dose that they were randomized to. We did not enroll children <3 years. We did not randomize by procedure type which could have confounded length of sedation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No